CLINICAL TRIAL: NCT01228708
Title: Effects of an Active Implementation of a Chronic Disease Management Programme for Patients With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Effects of an Active Implementation of a Guideline for Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Research Unit for General Practice, Aarhus University (Other); Ringkoebing-Skjern Municipality, Denmark. (Unknown); Region MidtJylland Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Active Implementation-FEAA
Record Dates: First submitted 2010-10-25; First posted 2010-10-26 (Estimated); Last update posted 2012-03-28 (Estimated); Status verified 2012-03

CONDITIONS: Implementation of a Chronic Disease Management Programme; COPD
Keywords: Implementation strategy; Chronic disease management programme; COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Intervention (Active Comparator): Patients from half the GP practices in Ringkoebing-Skjern municipality that participates in an active implementation of a guideline for COPD
  Interventions: Other: Active implementation of a guideline for chronic disease
- Control group (No Intervention): Patients from the half of the GP practice in Ringkoebing-Skjern that do not participate in the active implementation of a guideline for COPD. The GPs are however in postgraduate training groups with intervention groups GPs
- External control (No Intervention): Patients with GP practice in neighboring county Ikast-Brande where there have been no information or contact at all from the investigators

INTERVENTIONS:
Other: Active implementation of a guideline for chronic disease — Smoking cessation courses Remuneration to GPs for the planned follow-up and joint home visits Action card and sputum colour advice Webpage on "How to live with COPD" and the support the health system can provide Database with patients with COPD Feed-back from health centre to GPs, when patients have finished courses Fax from hospital to GPs, when patients with COPD is discharged Routines to recall patients for follow-ups Team audit, evaluate and adjust the strategies every 3rd month Joint home visit with GP and community nurse when a patient with COPD is discharged to plan future care Practice staff do part of follow-ups and monitoring Practice supervision with consultant in lung diseases Podcast with advice from specialists Guideline for COPD
  Arms: Intervention

SUMMARY:
Aims:

To design a proactive implementation strategy for a chronic-disease-management-programme.

To describe effects of the active implementation of a programme for COPD-patients measured on patient-related goals and use of health resources.

To describe stakeholders' evaluation of the implementation.

Materials and method:

An intervention study with 3000 COPD-patients cluster-randomized after a bloc-randomization of their GP-practice. 18 GP-practices in Ringkøbing-Skjern-Municipality are randomized to receive an active implementation or to an "as usual" group. A neighboring municipality acts as "sleeping" control. With data from registers and a questionnaire-survey the effect on COPD-patients self reported-health, evaluation of health system and changes in distribution of health resources is analyzed. How health professionals perceive the implementation and how it influences their conception, interactions and culture is illustrated by interviews with stakeholders.

We expect to see improved health related quality of life, enhanced evaluation of the health system and a more appropriate distribution of health resources in the intervention group.

DETAILED DESCRIPTION:
BACKGROUND:

Health systems will manage more and more people with chronic diseases as life-expectancy increases and treatment options improve. As the need for resources increases, it will be vital that a targeted strategy for health care to this growing group is developed so all are offered a professional and efficient treatment and that resources are used equitable. A proactive strategy will secure that not only acute needs of patients, but the need of the whole population is served.

AIM:

To describe the process of implementation and the effects of Central Denmark Region's chronic disease management programme for COPD-patients.

METHOD:

This is an intervention study, where approximately 3000 COPD-patients will be cluster-randomized after a bloc-randomization of their GP-practice. 15 GP-practices in Ringkøbing-Skjern Municipality will be randomized to receive the focused implementation or to an "as usual" group.

Approximately 4000 COPD patients from a neighboring municipality with a similar profile will be a control group without any active implementation in any GP-practice and any contamination between GP-practices will therefore be eliminated.

THE INTERVENTION:

A proactive implementation strategy for the chronic disease management programme will be designed based on the literature and methods which have proven effective in implementing new ways of working when different stakeholders and cultures are involved.

Core intervention elements: GP-practice visits and education with focus on registration of smoking status and offering of smoking cessation, stratification of COPD patients according to health level or disease status, written referral from GP to community initiatives and written feedback to GP, discharge notice to GP from hospital, home visit by GP or practice nurse together with community nurse to plan care with newly discharged frail patients,

With data from registers and a questionnaire-survey the effect on COPD-patients self reported health, evaluation of the health system and changes in the distribution of health resources will be analyzed. How the health professionals in hospital, community-care and in GP-practices perceive the implementation and how it influences their conception, interactions and culture will be illustrated in an interview-survey of stakeholders.

ELIGIBILITY:
Inclusion Criteria:

* People who live in either Ringkoebing-Skjern or Ikast-Brande municipalities and have a GP in the municipality and have been in hospital during the last 5 years with a lung related diagnosis or has redeemed a prescription for medication for lung related problems twice during the last year or has had at least two spirometries done during the last year.

Exclusion Criteria:

* People who do not fit the above inclusion criteria

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3021 (Actual)
Dates: Start 2009-08; Primary Completion 2010-10 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Changes in COPD-patients self reported-health, their evaluation of the health system and in the distribution of health resources. | 14 months

SECONDARY OUTCOMES:
Health professionals | 14 months
  How health professionals perceive the implementation and how it influences their conception, interactions and culture.

CONTACTS AND LOCATIONS:
Overall Officials: Margrethe IC Smidth, PT MSc, Principal Investigator — The Research Unit for General Practice Aarhus

REFERENCES:
- [Derived] Smidth M, Christensen MB, Fenger-Gron M, Olesen F, Vedsted P. The effect of an active implementation of a disease management programme for chronic obstructive pulmonary disease on healthcare utilization--a cluster-randomised controlled trial. BMC Health Serv Res. 2013 Oct 3;13:385. doi: 10.1186/1472-6963-13-385. PMID 24090189
- [Derived] Smidth M, Olesen F, Fenger-Gron M, Vedsted P. Patient-experienced effect of an active implementation of a disease management programme for COPD - a randomised trial. BMC Fam Pract. 2013 Oct 3;14:147. doi: 10.1186/1471-2296-14-147. PMID 24088417
- [Derived] Smidth M, Christensen MB, Olesen F, Vedsted P. Developing an active implementation model for a chronic disease management program. Int J Integr Care. 2013 Jun 17;13:e020. doi: 10.5334/ijic.994. Print 2013 Apr. PMID 23882169
- [Derived] Smidth M, Sokolowski I, Kaersvang L, Vedsted P. Developing an algorithm to identify people with Chronic Obstructive Pulmonary Disease (COPD) using administrative data. BMC Med Inform Decis Mak. 2012 May 22;12:38. doi: 10.1186/1472-6947-12-38. PMID 22616576